CLINICAL TRIAL: NCT04153032
Title: Comparative Evaluation of MEBO Ointment and Topical Diltiazem Ointment in the Treatment of Acute Anal Fissure: a Randomized Clinical Trial
Brief Title: Comparative Evaluation of MEBO Ointment and Topical Diltiazem Ointment in the Treatment of Acute Anal Fissure
Acronym: MEBO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Eman Sbaity, Instructor of Surgery, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2018-0547
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-07

CONDITIONS: Anal Fissure
Keywords: Anal fissure; MEBO; topical diltiazem; MEBO/Diltiazem combination
MeSH Terms: conditions — Fissure in Ano | interventions — Diltiazem

STUDY DESIGN:
Intervention Model Description: 1:1:1 randomized, controlled, parallel design
Who Masked: Investigator, Outcomes Assessor
Masking Description: The physician and the patient will not be blinded to the allocation, but the rest of the study team will be blinded. We will blind to allocation the physician who will assess for outcomes, and the research assistants who are collecting the data, data analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DTZ arm (Experimental): The first group of patients will apply MEBO ointment peri-anally 3 times daily for 6 weeks.
  Interventions: Drug: Mebo
- MEBO arm (Experimental): The second group of patients will apply topical DTZ ointment peri-anally 3 times daily for 6 weeks.
  Interventions: Drug: Diltiazem
- MEBO and DTZ arm (Experimental): The third group will apply a combination of MEBO and DTZ ointment peri-anally 3 times daily for 6 weeks. Those who fail therapy (meaning they report no pain improvement after two weeks of treatment) from either the MEBO or the Diltiazem arm will be switched to the combination arm. If they also fail to improve after two weeks on the treatment arm, then they will be offered surgery. If the patient refuses to switch to the combination arm and wishes to proceed to surgery immediately, then the patient will be directed to surgery.
  Interventions: Drug: Diltiazem; Drug: Mebo

INTERVENTIONS:
Drug: Diltiazem — DTZ is a calcium channel blocker for the treatment of chronic anal fissure
  Other Names: DTZ
  Arms: MEBO and DTZ arm; MEBO arm
Drug: Mebo — Moist exposed burn ointment (MEBO) is a tropical Chinese medicine composed of sesame oil and herbal plants that is clinically used for the treatment of burn wound.
  Arms: DTZ arm; MEBO and DTZ arm

SUMMARY:
No study to date has compared topical DTZ to MEBO ointment in the treatment of anal fissure. Therefore, the present study aims to compare the efficacy and safety of DTZ to MEBO in the treatment of acute anal fissure. The investigators propose to conduct a comparative randomized clinical study. In this study, the investigators will compare patients with acute anal fissure receiving MEBO ointment vs Topical DTZ ointment vs a combination of MEBO and DTZ ointment.

Hypothesis:

MEBO in combination with DTZ is more effective than DTZ or MEBO alone in the treatment of acute anal fissure.

DETAILED DESCRIPTION:
Trial Design: This trial is designed as a 1:1:1 randomized, controlled, parallel design. The primary endpoints are change in pain score and wound healing from baseline to 1 week from the study start date; secondary endpoints are change in pain score and wound healing at 6 and 10 weeks from the study start date, defecation strain score & the patient's global impression of improvement at 10 weeks.

Assessments & Visits: The patient will be assessed for pain, wound healing, strain during defecation, impression of improvement, & adverse events at weeks 1, 6 & 10 after the study start date. Trained resident or research assistant (RA) will administer the questionnaires on pain score, strain during defecation, & patient's global impression of improvement. During the follow-up visits, the average score for each of the pain & defecation strain scores will be taken for the 3 most recent days that the patient has defecated. The patient will be given a paper diary to record the pain score & strain score during defecation 3 days prior to the follow-up clinic visit.

Sample Size: The investigators will design this superiority trial as three-arm trials, where one arm is Diltiazem, second is MEBO, & last is a combination of both. Assuming that the pain score difference between both treatments will be 0.5 points with a 1-point standard deviation on the numeric rating scale (5 for DTZ & 3 for combination arm DTZ & MEBO), & using an alpha of 0.05 & a power of 80%, a sample size of 47 patients in each arm is needed. After accounting for a 30% loss to follow up, 61 patients will need to be recruited in each arm. The total number of patients to be recruited in the three arms is 183 patients.

Recruitment: At the American University of Beirut Medical Center, patients with acute anal fissure are treated at the outpatient center (private & outpatient clinics) of the hospital by all the general surgeons. The patients will be introduced to the study by their attending physician. If the patient agrees to participate, the RA (part of the research team) will approach & screen the patient according to the defined inclusion & exclusion criteria. If the patient is found eligible for the study, the RA will discuss the study & obtain his/her informed consent. The expected recruitment rate is 4 patients/week. The first 2 visits of the patient to the clinic at weeks 1 &6 from the start date of the study are part of clinical care & the patient will not be reimbursed for these visits. The last visit to the clinic that will take place at week 10 will be for follow-up as part of the research, so the patient and physician will be reimbursed for transportation and professional fees, respectively, by the research grant.

ASSIGNMENT OF INTERVENTIONS

Sequence Generation: Participants will be randomly assigned to their treatment in a 1:1:1 ratio, according to a computer-generated schedule, stratified by type of treatment (MEBO or DTZ), using permuted blocks of variable sizes.

Allocation Concealment Mechanism: Random sequence generation will be selected by CRI biostatistician using computer software. The CRI person will hold details of the blocking & block sizes in a separate document unavailable to those involved in the study so ensure allocation concealment. The CRI person will not share the treatment intervention with study personnel until baseline characteristics are collected, & the patient is recruited into the trial. The physician will contact the CRI biostatistician & receive treatment allocation, so he/she can prescribe the ointment to which the patient is randomized to.

Implementation: The CRI biostatistician, who is not involved in this study, will generate the randomization sequence & keep hold of it. The patient will be recruited & consented without any knowledge about their allocation arm. The allocation will be revealed only to the physician to administer the treatment.

Blinding: The physician & the patient will not be blinded to the allocation, but the rest of the study team will be blinded. It is difficult to blind the physician or patient because of the characteristic smell of MEBO that is easily recognizable. Also blinded to allocation is the physician who will assess for outcomes, the RA who are collecting the data, & data analyst.

DATA COLLECTION, MANAGEMENT, & ANALYSIS

Data Collection Methods: Data on basic demographics of the study subjects, relevant risk factors, confounders, & indication for the type of treatment will be collected at baseline using protocol-specific standardized case report forms (CRF). The CRF will be completed by the RA directly from patients, following informed consent & prior to the administration of treatment. The different sections of that data will be collected at the different points in time of the study by questionnaires administered by the study RA to the patient. Evaluators are requested to fill immediately a case report form each time an outcome evaluation on a study subject is performed. These forms will be handed in the same setting to the RA who will take care of storing them. To improve retention & compliance to the study, the investigators will contact the patient ahead of time, & help schedule their clinic visits on time to collect the outcomes. When a patient fails to comply with the follow-up exams, the investigators will collect applicable data on the phone (Appendix C). For those who drop from the study, the investigators will analyze their basic demographic & disease data to determine whether or not those are similar to those who stayed on the study.

Data Management: The RA will enter the data from the CRFs on the study data excel sheet within 1 week of its collection. The data will be manually entered twice & independently by the RA & another member of the study team. Data will be entered as the actual numeric values or categorical variables, initially. In the end, the statistician will code all the data in preparation for analysis. The principal investigator (PI) will perform spot checks on the data & will review weekly all the CRF & assessment collection sheets performed within each week. At AUBMC, data will be stored on the AUB intranet server on the PI's computer. All research members will have access to the data. The Case Report Forms will be stored in a locked cabinet in the PI office 3 years following the publication of study results. The investigators will provide an SOP detailing data management procedure to ensure consistency in case of a change in the study members. Audits will be performed monthly on 20% of the charts.

Statistical Methods: the investigators will compare the three arms for the primary, secondary, & exploratory outcomes. The investigators will use the chi-square or Fischer exact test if the expected count of any of the outcomes is less than 5 per cell for analysis of the incidence of categorical outcomes (like wound healing). The investigators will use the independent t-test for analysis of the continuous outcomes (like pain score, defecation strain score, Patient's Global Impression of Improvement). The investigators will calculate relative risk with corresponding 95% confidence intervals to compare the incidence of the categorical outcomes while reporting a difference in means for the continuous outcomes. SPSS version 20 will be used to conduct the analysis. A 2 sided p-value will be set at 5%. The univariate analysis will be performed separately for the two primary outcomes & the three secondary outcomes at weeks 1, 6 & 10. Multivariate analysis for change in pain score & wound healing will be performed using linear regression and logistic regression respectively, controlling for age, gender, duration of the anal fissure since presentation, analgesic medications intake (only with pain score), defecation strain score. The investigators will perform both ITT & PP analysis for all outcome measures. The ITT analysis will include all patients randomized per arm. In case of failure of treatment in one of the arms, those who will switch to another arm will be still analyzed as part of the arm initially randomized to. Multiple imputation methods will be used to handle missing data. To assess the effect of missing data on the analysis, sensitivity analyses will be performed. The study biostatistician will perform the best case scenario, worst-case scenario, & group averages. The investigators will assess the baseline characteristics of those who will be lost to follow up, which would help understand what were the potential outcomes.

DATA MONITORING

Data Monitoring Committee: The DMC will be independent of the PI & funders of the trial & composed of a surgeon, an internist, a nurse, a biostatistician, & a representative from the patient advocacy office at AUBMC. The internist will have a clinical research background. The nurse is chosen from the inpatient floors, to make sure that there is no interaction with study subjects. All members should not have any conflict of interest related to the study. The DMC will be chaired by the internist, who has to keep a record of the meetings & recommendations for future reference. Since this is an investigator-initiated trial, the PI will appoint the DMC members. The DMC will meet every other month, at times of scheduled interim analysis, & upon conclusion of the study. The primary role of the DMC is to review accumulating data & alert the steering committee if there are alarming rates of side effects (SE) in any arm of the trial. This committee doesn't have executive power to stop the trial or modify treatment. The committee will report results to the PI. In addition, the DMC will keep track of the accrual rate.

Interim Analysis: The interim analysis will be done 3 times throughout the study; upon recruiting quarter, two-quarters, & three-quarters of the study population. The study biostatistician who is blind to the treatment allocations will conduct the interim analysis & will use the O'Brien Fleming stopping rules. The study biostatistician will report the results of the interim analysis to the DMC confidentially. At each interim-analysis interpretation, the DMC will alert the PI if one arm is found to be beyond doubt either more beneficial or more harmful than the other arm. The PI will take into consideration the results of the interim analysis, opinion of the DMC, & various important factors to decide upon the fate of the trial. The chairperson of the DMC will monitor the ClinicalTrials.gov website for registration of new trials & for newly reported results from trials addressing the similar questions as this trial.

Harms: The adverse effects can be part of the outcome measures detailed earlier in the protocol or other not specified SEs. Either way, any SE will be reported & the subject will be managed according to the standard of care or the preference of the treating physician. In case any adverse effects arise outside scheduled follow-up time, the patient will be seen by the treating physician in an extra add-on visit. Those who fail (meaning those who do not report any pain improvement after two weeks of treatment) from either the MEBO or the Diltiazem arm will be switched to the combination arm. If these patients also fail to improve after 2 weeks on the combination arm, then the patient will be offered surgery. If the patient refuses to switch to the combination arm & wishes to proceed to surgery immediately, then the patient will be directed to surgery. In case of failure of the treatment, which is after 6 weeks of treatment, the patient will undergo surgery. The patient may also undergo surgery in case he/she decides to stop medical therapy during the treatment period & proceed to surgery. There is no standard for the risk of failure of topical therapy to necessitate surgery. Hence, the risk of failure cannot be evaluated with the use of MEBO.

The primary physician who is treating the patient will be responsible for the management of the SEs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years and above.

  * Subjects with 3 months (90 days) or less history of painful anal fissure (AF), prior to screening, where AF-related pain-associated with, or following, defecation is experienced at least twice a week during the symptomatic phase, with pain scores at an average of ≥ 3 on an 11-point NRS (Numerical Rating Scale, range 0-10 where 0 = no pain and 10 = worst pain imaginable).
  * Subjects with an average of ≥4 on an 11-point NRS during the screening phase for worst anal pain associated with, or following, defecation for the most recent 3 days on which the subject has defecated.
  * Subjects with evidence of a radial fissure, with induration at the edges, seen on anal examination.
  * Willing to stop all other concomitant topical preparations applied perianally prior to commencing study treatment, and throughout the study. There will be a "washout" period of at least 2 weeks prior to commencing the study for subjects who were using other concomitant topical preparations applied perianally.
  * Able to give consent

Exclusion Criteria:

* Subjects unwilling to be examined for AF.
* Subjects who have undergone the following procedures:

  * Lateral sphincterotomy or anal stretch or other previous surgery involving the anal canal or perianal region (hemorrhoidectomy, anal fistula surgery).
  * Incision of perianal abcess.
* Subjects who have had sub-fissure injection of botulinum toxin within 6 months period prior to screening, or have used glyceryl trinitrate (GTN) ointment for >1 week in the 4 weeks prior to the screening visit.
* Subjects with AF associated with other conditions (drug-induced [e.g. nicorandil], trauma, HIV infection, fistula-in-ano, inflammatory bowel disease, perianal sepsis or malignancy).
* Subjects with cardiovascular disease
* Subjects with known hypersensitivity to DTZ or the ingredients of MEBO (Sesame oil)
* Subjects taking medications prohibited by the protocol.
* Subjects who have taken experimental agents must have been discontinued at least 8 weeks prior to screening, or for a period equivalent to 5 half-lives (t1/2) of the agents.
* Subjects who have the following gastrointestinal disorders:

  * Inflammatory bowel disease.
  * Chronic faecal incontinence.
  * History of radiation therapy to the pelvis.
  * Fixed anal stenosis/fibrosis.
* Subjects with major psychiatric (including drug or alcohol abusers), or haematological illness. (diseases of the vascular system; source: )Subjects with planned elective or other treatment requiring hospitalization, during the study, booked before entry into the study.
* Subjects who will be unavailable for the duration of the trial, likely to be noncompliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason.
* Patients who are taking oral therapy for anal fissure will also be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Score | Baseline to 1 week from the start date of the study
  Pain is evaluated through the Numerical Rating Scale, range 0-10 where 0 = no pain and 10 = worst pain imaginable
Wound Healing | At 1 week from that start date of the study
  Wound healing is assessed through physical examination: digital rectal examination is not done in case of painful anal fissure. Assessment for wound healing will be performed by the treating physician of the patient. The patient will be asked to strain to make the anal fissure more visible. If it is difficult to see on physical examination, digital rectal exam is done carefully. The degree of healing will be reported as none, partial or complete.

SECONDARY OUTCOMES:
Change in Pain Score | At 6 and 10 weeks from the start date of the study
  Pain is evaluated through the Numerical Rating Scale, range 0-10 where 0 = no pain and 10 = worst pain imaginable
Wound Healing | At 6 and 10 weeks from the start date of the study
  Wound healing is assessed through physical examination: digital rectal examination is not done in case of painful anal fissure. Assessment for wound healing will be performed by the treating physician of the patient. The patient will be asked to strain to make the anal fissure more visible. If it is difficult to see on physical examination, digital rectal exam is done carefully.
Defecation Strain Score | At 1 week, 6 weeks, and 10 weeks from that start date of the study
  Level of strain during defecation is graded on a four-point scale: serious strain was scored as 3, moderate strain as 2, mild strain as 1, and defecation without strain as 0
Global Impression of Improvement | At 1 week, 6 weeks, and 10 weeks from that start date of the study
  The patient's global impression of improvement will be measured on a 7-point Likert scale where 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse.

OTHER OUTCOMES:
Incidence of Treatment-Related Adverse Events | At 1 week, 6 weeks, and 10 weeks from that start date of the study
  Incidence of Headache, Itching, Dizziness, Hypersensitivity reactions or Critical Change in Vital Signs.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Sbaity, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hadianamrei R. Topical diltiazem in management of chronic anal fissure: a review of the literature. Clinical Investigation. 2014;4(10):923-34.
- [Background] Sailer M, Bussen D, Debus ES, Fuchs KH, Thiede A. Quality of life in patients with benign anorectal disorders. Br J Surg. 1998 Dec;85(12):1716-9. doi: 10.1046/j.1365-2168.1998.00958.x. PMID 9876082
- [Background] Ram E, Alper D, Stein GY, Bramnik Z, Dreznik Z. Internal anal sphincter function following lateral internal sphincterotomy for anal fissure: a long-term manometric study. Ann Surg. 2005 Aug;242(2):208-11. doi: 10.1097/01.sla.0000171036.39886.fa. PMID 16041211
- [Background] Herzig DO, Lu KC. Anal fissure. Surg Clin North Am. 2010 Feb;90(1):33-44, Table of Contents. doi: 10.1016/j.suc.2009.09.002. PMID 20109631
- [Background] Li W, Ma Y, Yang Q, Pan Y, Meng Q. Moist exposed burn ointment for treating pressure ulcers: A multicenter randomized controlled trial. Medicine (Baltimore). 2017 Jul;96(29):e7582. doi: 10.1097/MD.0000000000007582. PMID 28723796
- [Background] Hirsch T, Ashkar W, Schumacher O, Steinstraesser L, Ingianni G, Cedidi CC. Moist Exposed Burn Ointment (MEBO) in partial thickness burns - a randomized, comparative open mono-center study on the efficacy of dermaheal (MEBO) ointment on thermal 2nd degree burns compared to conventional therapy. Eur J Med Res. 2008 Nov 24;13(11):505-10. PMID 19073386
- [Background] Ang ES, Lee ST, Gan CS, See P, Chan YH, Ng LH, Machin D. The role of alternative therapy in the management of partial thickness burns of the face--experience with the use of moist exposed burn ointment (MEBO) compared with silver sulphadiazine. Ann Acad Med Singap. 2000 Jan;29(1):7-10. PMID 10748957
- [Background] National Institute for Health and Care Excellence. Chronic anal fissure: 2% topical diltiazem hydrochloride. Evidence Summary. Manchester: 2013.
- [Background] Schochet E, Khubchandani I. Pathophysiology of Chronic Anal Fissure: Current Understanding and Clinical Applications. Societa Italiana di Chirurgia ColoRettale. 2007;15:130-5.
- [Background] Bansal AR, Yadav PK, Godara R, Pal N, Tripura R, Jaikaran. Comparative evaluation of 0.2% glyceryl trinitrate vs. 2% diltiazem ointment in treatment of chronic anal fissure treatment - a randomized trial. Hellenic Journal of Surgery. 2016;88(1):25-30.
- [Background] Steele SR, Madoff RD. Systematic review: the treatment of anal fissure. Aliment Pharmacol Ther. 2006 Jul 15;24(2):247-57. doi: 10.1111/j.1365-2036.2006.02990.x. PMID 16842451
- [Background] Antropoli C, Perrotti P, Rubino M, Martino A, De Stefano G, Migliore G, Antropoli M, Piazza P. Nifedipine for local use in conservative treatment of anal fissures: preliminary results of a multicenter study. Dis Colon Rectum. 1999 Aug;42(8):1011-5. doi: 10.1007/BF02236693. PMID 10458123
- [Background] Collins EE, Lund JN. A review of chronic anal fissure management. Tech Coloproctol. 2007 Sep;11(3):209-23. doi: 10.1007/s10151-007-0355-9. Epub 2007 Aug 3. PMID 17676270
- [Background] Amir H, Tibi Y, Groutz A, Amit A, Azem F. Unpredicted gender preference of obstetricians and gynecologists by Muslim Israeli-Arab women. Patient Educ Couns. 2012 Feb;86(2):259-63. doi: 10.1016/j.pec.2011.05.016. Epub 2011 Jun 16. PMID 21680130
- [Background] Medhi B, Rao RS, Prakash A, Prakash O, Kaman L, Pandhi P. Recent advances in the pharmacotherapy of chronic anal fissure: an update. Asian J Surg. 2008 Jul;31(3):154-63. doi: 10.1016/S1015-9584(08)60078-0. PMID 18658016
- [Background] Medhi B, Prakash A, Upadhyay S, Xess D, Yadav TD, Kaman L. Comparison of observational and controlled clinical trials of diltiazem in the treatment of chronic anal fissure. Indian J Surg. 2011 Dec;73(6):427-31. doi: 10.1007/s12262-011-0340-4. Epub 2011 Oct 18. PMID 23204700
- [Background] Tsunoda A, Kashiwagura Y, Hirose K, Sasaki T, Kano N. Quality of life in patients with chronic anal fissure after topical treatment with diltiazem. World J Gastrointest Surg. 2012 Nov 27;4(11):251-5. doi: 10.4240/wjgs.v4.i11.251. PMID 23494072
- [Background] Stewart DB Sr, Gaertner W, Glasgow S, Migaly J, Feingold D, Steele SR. Clinical Practice Guideline for the Management of Anal Fissures. Dis Colon Rectum. 2017 Jan;60(1):7-14. doi: 10.1097/DCR.0000000000000735. No abstract available. PMID 27926552
- [Background] Katsinelos P, Kountouras J, Paroutoglou G, Beltsis A, Chatzimavroudis G, Zavos C, Katsinelos T, Papaziogas B. Aggressive treatment of acute anal fissure with 0.5% nifedipine ointment prevents its evolution to chronicity. World J Gastroenterol. 2006 Oct 14;12(38):6203-6. doi: 10.3748/wjg.v12.i38.6203. PMID 17036396
- [Background] Guo-Lin H, Zhong-shen L. Experience with MEBO in Treating 42 Cases of Anal Fissure. The Chinese Journal of Burns Wounds and Surface Ulcers. 2001(2).
- [Background] Zhong-gui C, Jun Z, Ze-zi A. Analysis of the efficacy of MEBO in treating 51 cases of anal fissure. The Chinese Journal of Burns Wounds & Surface Ulcers 2004(3).
- [Background] Patankar R, Mishra A. A prospective non-comparative study to assess the effectiveness and safety of combination laxative therapy containing milk of magnesia, liquid paraffin and sodium picosulphate (Cremaffin-Plus®) in the management of constipation in patients with anal fissure/hemorrhoids/obstructive defecation syndrome. International Surgery Journal. 2017;4(12).
- [Background] Srikrishna S, Robinson D, Cardozo L. Validation of the Patient Global Impression of Improvement (PGI-I) for urogenital prolapse. Int Urogynecol J. 2010 May;21(5):523-8. doi: 10.1007/s00192-009-1069-5. Epub 2009 Dec 15. PMID 20013110
- [Derived] El Charif MH, Doughan S, Kredly R, Kassas S, Azab R, Sbaity E. MEBO versus topical Diltiazem versus a combination of both ointments in the treatment of acute anal fissure: a randomized clinical trial protocol. BMC Complement Med Ther. 2021 Feb 24;21(1):75. doi: 10.1186/s12906-021-03227-z. PMID 33627111